CLINICAL TRIAL: NCT00939341
Title: Real Life Effectiveness of Symbicort Maintenance and Reliever Therapy (SMART) in Asthma Patients Across Asia: SMARTASIA
Brief Title: Study to Investigate Real Life Effectiveness of Symbicort Maintenance and Reliever Therapy in Asthma Patients Across Asia
Acronym: SMARTASIA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5890L00035
Record Dates: First submitted 2009-07-13; First posted 2009-07-15 (Estimated); Results first posted 2011-11-28 (Estimated); Last update posted 2012-01-16 (Estimated); Status verified 2012-01

CONDITIONS: Asthma
Keywords: Symbicort SMART
MeSH Terms: conditions — Asthma | interventions — Budesonide, Formoterol Fumarate Drug Combination; Budesonide; Formoterol Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Symbicort Turbuhaler 160/4.5 µg delivered dose
  Interventions: Drug: Symbicort (Budesonide/Formoterol)

INTERVENTIONS:
Drug: Symbicort (Budesonide/Formoterol) — Turbuhaler 160/4.5 µg delivered dose, twice daily (one inhalation in the morning and one inhalation in the evening) and as need (prn) in response to symptoms
  Other Names: Symbicort

SUMMARY:
The purpose of this study is to compare whether Symbicort Maintenance & Reliever Therapy (SMART) is more effective in uncontrolled asthmatic patients than their current therapy in a real life situation.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed informed consent
* Asthma diagnosis at least 6 months before visit 1 of study
* Patients who have reversible airway obstruction continuous asthma treatment except Symbicort at least within 4 weeks before visit 1 of study

Exclusion Criteria:

* Known or suspected allergy to active ingredients of study medication or excipients
* Use of oral, rectal or parenteral glucocorticosteroids 30 days before visit 1 of study
* Smoking, current or previous with a smoking history of ≥ 10 pack years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 862 (Actual)
Dates: Start 2009-07; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guy Yeoman, MD, Study Director — AstraZeneca
Locations (35):
- China (13):
  - Research Site, Guangzhou, Guangdong
  - Research Site, Zheng Ahou, Henan
  - Research Site, Wuhan, Hubei
  - Research Site, Changsha, Hunan
  - Research Site, Qingdao, Shandong
  - Research Site, Shanghai, Shanghai Municipality
  - Research Site, Beijing
  - Research Site, Chengdu
  - Research Site, Fuzhou
  - Research Site, Hangzhou
  - Research Site, Nanjing
  - Research Site, Shenyang
  - Research Site, Zhengzhou
- India (10):
  - Research Site, Hyderabad, Andhra Pradesh
  - Research Site, Ahmedabad, Gujarat
  - Research Site, Bangalore, Karnataka
  - Research Site, Bengaluru, Karnataka
  - Research Site, Indore, Madhya Pradesh
  - Research Site, Mumbai, Maharashtra
  - Research Site, Chennai, Tamil Nadu
  - Research Site, Coimbatore, Tamil Nadu
  - Research Site, Lucknow, Uttar Pradesh
  - Research Site, Noida, Uttar Pradesh
- Indonesia (2):
  - Research Site, Jakarta, DKI Jakarta
  - Research Site, Surabaya, East Java
- Taiwan (6):
  - Research Site, Chiayi City
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Taipei
  - Research Site, Taoyuan
  - Research Site, Taoyuan District
- Thailand (4):
  - Research Site, Bangkok, Bangkok
  - Research Site, Pathumwan, Bangkok
  - Research Site, Pathum Thani, Changwat Pathum Thani
  - Research Site, Nakhonratchasima, Naimuang

REFERENCES:
- [Derived] Lin J, Tang Y, Xiu Q, Kang J, Cai S, Huang K, Itoh Y, Ling X, Zhong N. Real-life effectiveness of budesonide/formoterol therapy in asthma: A subanalysis of the SMARTASIA study. Allergy Asthma Proc. 2016 Jan-Feb;37(1):27-34. doi: 10.2500/aap.2016.37.3910. PMID 26831844
- [Derived] Zhong N, Lin J, Mehta P, Ngamjanyaporn P, Wu TC, Yunus F. Real-life effectiveness of budesonide/formoterol maintenance and reliever therapy in asthma patients across Asia: SMARTASIA study. BMC Pulm Med. 2013 Apr 4;13:22. doi: 10.1186/1471-2466-13-22. PMID 23557023

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1022 asthma patients were enrolled at 51 sites in 5 Asian countries: China (21 sites), India (12 sites), Indonesia (3 sites), Thailand (6 sites) and Taiwan (9 sites) during the period July 2009 to August 2010. Of the 1022 enrolled, 862 participants entered into a 12-week treatment with the investigational drug.
Pre-assignment Details: The study consisted of an initial screening visit followed by a 2-week run-in period before a 12-week treatment with investigational drug.
Groups:
- Symbicort Turbuhaler: 160/4.5 µg delivered dose
Period: Overall Study
Arm/Group | Symbicort Turbuhaler
Started | 862 (1022 participants were enrolled. There were 160 screen failures, 862 proceeded to treatment period.)
Completed | 796 (862 participants entered into the 12-week treatment,66 discontinued, 796 completed the treatment.)
Not Completed | 66
Not completed — Adverse Event | 15
Not completed — Pregnancy | 1
Not completed — Lost to Follow-up | 23
Not completed — Withdrawal by Subject | 13
Not completed — Protocol Violation | 6
Not completed — Incorrect enrolment | 8

BASELINE CHARACTERISTICS:
Arm/Group | Symbicort Turbuhaler
Number analyzed (Participants) | 862
Age Continuous [Mean (Standard Deviation); unit: Years]
  All Participants | 13.7 (44.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 455
  Male | 407

OUTCOME MEASURES:

1. Primary Outcome: Change in Asthma Control Questionnaire (ACQ(5)) Score From Baseline at a Regional Level
Description: Participants' levels of asthma control were scored on a 7-point Likert scale from 0 to 6, whereby 0 represents good control and 6 represents poor control of asthma. The regional mean change of overall ACQ(5) score were calculated as change from baseline (Week 0) to the average during the treatment period (mean of scores at Week 4, Week 8, Week 12).
Time Frame: Baseline and 12 weeks
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Symbicort Turbuhaler
Number analyzed (Participants) | 841
Units on a scale | -0.58 (-0.64) [-0.64 to -0.51]

2. Secondary Outcome: Change in ACQ(5) Score From Baseline at Country Level (China)
Description: as for outcome 1
Time Frame: Baseline and 12 weeks
Population: This outcome measure is reported at individual country level only, and therefore the number of patients analyzed are less than reported in participant flow, which captures the total patients in the region.
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Symbicort Turbuhaler
Number analyzed (Participants) | 386
Units on a scale | -0.58 (-0.67) [-0.67 to -0.49]

3. Secondary Outcome: Change in Overall ACQ(5) Score From Baseline at Country Level (India)
Description: as for outcome 1
Time Frame: Baseline and 12 weeks
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Symbicort Turbuhaler
Number analyzed (Participants) | 159
Units on a scale | -0.74 (-0.92) [-0.92 to -0.57]

4. Secondary Outcome: Change in Overall ACQ(5) Score From Baseline at Country Level (Indonesia)
Description: as for outcome 1
Time Frame: Baseline and 12 weeks
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Symbicort Turbuhaler
Number analyzed (Participants) | 61
Units on a scale | -1.18 (-1.40) [-1.40 to -0.95]

5. Secondary Outcome: Change in Overall ACQ(5) Score From Baseline at Country Level (Taiwan)
Description: as for outcome 1
Time Frame: Baseline and 12 weeks
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Symbicort Turbuhaler
Number analyzed (Participants) | 100
Units on a scale | -0.22 (-0.38) [-0.38 to -0.06]

6. Secondary Outcome: Change in Overall ACQ(5) Score From Baseline at Country Level (Thailand)
Description: as for outcome 1
Time Frame: Baseline and 12 weeks
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Symbicort Turbuhaler
Number analyzed (Participants) | 128
Units on a scale | -0.36 (-0.48) [-0.48 to -0.23]

7. Secondary Outcome: Change in Asthma Quality of Life Questionnaire, Standardized Version (AQLQ (S)) Overall Scores From Baseline
Description: Participants' QOL were scored on a scale of decreasing QOL impairment from 1 to 7, in which 1 = maximum impairment. The change in overall mean AQLQ(S) score from baseline were calculated as change from baseline (Week 0) to the average during the treatment period (mean of scores at Week 4, Week 8, Week 12)
Time Frame: Baseline and 12 weeks
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Symbicort Turbuhaler
Number analyzed (Participants) | 842
Units on a scale | 0.70 (0.64) [0.64 to 0.76]

8. Secondary Outcome: Change in AQLQ (S) Domain (Symptom) Scores From Baseline
Description: Participants' QOL were scored on a scale of decreasing QOL impairment from 1 to 7, in which 1 = maximum impairment. The change in overall mean AQLQ(S) symptom score were calculated as change from baseline (Week 0) to the average during the treatment period (mean of scores at Week 4, Week 8, Week 12).
Time Frame: Baseline and 12 weeks
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Symbicort Turbuhaler
Number analyzed (Participants) | 842
Units on a scale | 0.77 (0.70) [0.70 to 0.84]

9. Secondary Outcome: Change in AQLQ (S) Domain (Activity Limitation) Scores From Baseline
Description: Participants' QOL were scored on a scale of decreasing QOL impairment from 1 to 7, in which 1 = maximum impairment. The change in overall mean AQLQ(S) symptom score from baseline were calculated as change from baseline (Week 0) to the average during the treatment period (mean of scores at Week 4, Week 8, Week 12)
Time Frame: Baseline and 12 weeks
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Symbicort Turbuhaler
Number analyzed (Participants) | 842
Units on a scale | 0.59 (0.53) [0.53 to 0.65]

10. Secondary Outcome: Change in AQLQ (S) Domain (Emotion Function) Scores From Baseline
Description: Participants' emotional functions were scored on a scale of decreasing impairment to emotional function from 1 to 7, in which 1 = maximum impairment. The change in overall mean AQLQ(S) emotion function score were calculated as change from baseline (Week 0) to the treatment period (mean of the scores at Week 4, Week 8, Week 12)
Time Frame: Baseline and 12 weeks
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Symbicort Turbuhaler
Number analyzed (Participants) | 842
Units on a scale | 0.77 (0.70) [0.70 to 0.84]

11. Secondary Outcome: Change in AQLQ (S) Domain (Environmental Stimuli) Scores From Baseline
Description: Participants ' responses to environmental stimuli were scored on a scale of decreasing response to environmental stimuli from 1 to 7, in which 1 = maximum response. The change in overall mean AQLQ(S) score were calculated as change from baseline (Week 0) to the average during the treatment period (mean of scores at Week 4, Week 8, Week 12)
Time Frame: Baseline and 12 weeks
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Symbicort Turbuhaler
Number analyzed (Participants) | 842
Units on a scale | 0.67 (0.60) [0.60 to 0.74]

12. Secondary Outcome: Study Medication Use (Maintenance and Reliever) in Diary Cards - Change in As-needed Day-time Reliever Medication From run-in Period
Description: Change in the number of as-needed day-time inhalations of medication, defined as the difference in mean value of all available data obtained during treatment period and mean value in run-in period.
Time Frame: Baseline and 12 weeks
Measure: Mean (95% Confidence Interval); unit: Number of inhalations
Arm/Group | Symbicort Turbuhaler
Number analyzed (Participants) | 841
Number of inhalations | -0.30 (-0.36) [-0.36 to -0.23]

13. Secondary Outcome: Study Medication Use (Maintenance and Reliever) in Diary Cards - Change in As-needed Night-time Reliever Medication From run-in Period
Description: Change in the number of as-needed night-time inhalations of medication, calculated as difference in mean value of all available data obtained during treatment period and mean value in run-in period.
Time Frame: Baseline and 12 weeks
Measure: Mean (95% Confidence Interval); unit: Number of inhalations
Arm/Group | Symbicort Turbuhaler
Number analyzed (Participants) | 852
Number of inhalations | -0.30 (-0.35) [-0.35 to -0.24]

14. Secondary Outcome: Study Medication Use (Maintenance and Reliever) in Diary Cards - Total Number of Inhalations of Symbicort® 160µg/4.5µg Per Day During Treatment Period
Description: Total number of inhalations of Symbicort® 160µg/4.5µg per day during treatment period, defined as the sum of maintenance medication and as-needed medication during night and day time
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: Number of inhalations
Arm/Group | Symbicort Turbuhaler
Number analyzed (Participants) | 858
Number of inhalations | 2.51 (0.93)

15. Secondary Outcome: Study Medication Use (Maintenance and Reliever) in Diary Cards - Percentage of Days During Treatment Period Participants Used ≥ 3 Inhalations of Symbicort® 160µg/4.5µg in a Day
Description: The mean percentage of days during treatment period participants used ≥ 3 inhalations of Symbicort® 160µg/4.5µg in a day
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | Symbicort Turbuhaler
Number analyzed (Participants) | 858
Percentage of days | 28.25 (33.03)

16. Secondary Outcome: Study Medication Use (Maintenance and Reliever) in Diary Cards - Percentage of Days During Treatment Period Participants Used ≥ 5 Inhalations of of Symbicort® 160µg/4.5µg in a Day
Description: The mean percentage of days during treatment period participants used ≥ 5 inhalations of Symbicort® 160µg/4.5µg in a day
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | Symbicort Turbuhaler
Number analyzed (Participants) | 858
Percentage of days | 6.21 (16.17)

17. Secondary Outcome: Study Medication Use (Maintenance and Reliever) in Diary Cards - Percentage of Days During Treatment Period Participants Used ≥ 9 Inhalations of Symbicort® 160µg/4.5µg in a Day
Description: The mean percentage of days during treatment period participants used ≥ 9 inhalations of Symbicort® 160µg/4.5µg in a day
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | Symbicort Turbuhaler
Number analyzed (Participants) | 858
Percentage of days | 0.19 (1.92)

ADVERSE EVENTS:
Arm/Group | Symbicort Turbuhaler
Serious Adverse Events (participants affected / at risk) | 12/862
Other Adverse Events (participants affected / at risk) | 0/862
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Symbicort Turbuhaler (N=862)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2
Headache (Nervous system disorders) | 1
Cerebral Infarction (Nervous system disorders) | 1
Myocardial Infarction (Cardiac disorders) | 1
Nasal Polyps (Respiratory, thoracic and mediastinal disorders) | 1
Post procedural haemorrhage (Surgical and medical procedures) | 1
Pneumonia (Infections and infestations) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Renal Cysts (Renal and urinary disorders) | 1
Appendicitis (Infections and infestations) | 1
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Breast Cancer (Reproductive system and breast disorders) | 1
Atrioventricular block complete (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
The design of the study does not allow for any conclusion regarding the effect of Symbicort SMART, it being a within-group comparison

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No